CLINICAL TRIAL: NCT00544167
Title: A Pilot Study of Adjuvant Doxorubicin and Cyclophosphamide Followed by Paclitaxel Plus Sorafenib in Women With Node Positive or High-Risk Early Stage Breast Cancer
Brief Title: Adjuvant Doxorubicin/Cyclophosphamide and Paclitaxel Plus Sorafenib Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 112
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Early Stage; High Risk; Node Positive; Doxorubicin; Cyclophosphamide; Paclitaxel; Sorafenib
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All patients received doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 (AC) both administered intravenously day 1 every 3 weeks for four cycles, followed by paclitaxel 175 mg/m2 intravenously day 1 every 3 weeks for four cycles or 80 mg/m2 for twelve weeks (physician discretion), combined with sorafenib 400 mg orally twice daily. Sorafenib was held during radiation therapy where indicated and resumed once completed. Sorafenib was continued for a total of 12 months and in combination with adjuvant hormonal therapy where indicated.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Sorafenib

INTERVENTIONS:
Drug: Doxorubicin
  Other Names: Adriamycin
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Paclitaxel
  Other Names: Taxol
Drug: Sorafenib
  Other Names: Nexavar

SUMMARY:
Sorafenib is being looked at in a number of solid tumor settings including breast cancer. This trial is designed as a pilot study to assess the safety and tolerability of a novel oral agent in combination with standard chemotherapy in the treatment of early stage node positive or otherwise high-risk breast cancer. If this should prove to be a tolerable regimen for patients, this would provide rationale for further studies in a larger randomized fashion.

DETAILED DESCRIPTION:
Primary Objectives The primary objective is to assess the safety and tolerability of doxorubicin / cyclophosphamide followed by paclitaxel in combination with sorafenib in patients with early stage node positive or otherwise high-risk breast cancer.

Secondary Objectives The secondary objectives are to assess activity in the form of recurrence-free-interval, distant recurrence-free interval,and overall survival in this pilot study of doxorubicin / cyclophosphamide followed by paclitaxel in combination with sorafenib in patients with early stage node positive or otherwise high-risk breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed breast cancer with an interval between definitive surgery that includes axillary lymph node involvement assessment and initiation of study treatment of less than or equal to 84 days.
* Definitive surgery - either mastectomy with axillary node involvement assessment, or breast conserving surgery with axillary node assessment. Margins of resected specimen must be free of invasive disease and/or ductal carcinoma in situ (DCIS).
* Stage I, II, IIIA, and IIIC (T1-3, N3a only). Patients must be either lymph node positive or high-risk node negative.
* Age > 18 years.
* ECOG performance status 0 or 1.
* Normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF) by Echocardiography or MUGA scan and electrocardiogram (ECG) within 35 days prior to initiation of study treatment.
* Patients must have adequate bone marrow function
* Patients must have normal liver function (
* Serum creatinine <= 2mg/dl
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored.

Exclusion Criteria:

* Prior systemic anticancer therapy for breast cancer (immunotherapy, chemotherapy, hormonal therapy).
* Patients with HER2 positive breast cancer as determined by FISH or IHC3+ standing are ineligible for this trial.
* Prior anthracycline or taxane therapy.
* Prior radiation therapy for breast cancer.
* Bilateral invasive disease.
* Pre-existing motor or sensory neurotoxicity of a severity ≥ 2 by NCI CTCAE v 3.0 criteria.
* Cardiac disease that includes: myocardial infarction; angina, congestive heart failure, arrhythmia; valvular heart disease; cardiomegaly on chest imaging or ventricular hypertrophy on ECG - unless the LVEF is within normal range for the institution; patients with poorly controlled hypertension (defined as systolic blood pressure > 150 and /or diastolic blood pressure > 100 mmHg on antihypertensive medications); patients who receive medications for angina, arrhythmias, or congestive heart failure.
* Current therapy with raloxifene, tamoxifen or other selective estrogen receptor modulator
* Concurrent treatment with ovarian hormonal replacement therapy.
* History of prior malignancy within 5 years with the exception of skin cancer or cervical carcinoma in situ.
* Women who are pregnant (positive pregnancy test) or breast feeding. Subjects of childbearing potential must use effective birth control measures during treatment.
* Treatment with a non-approved or investigational drug within 30 days before day 1 of trial treatment.
* Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Thrombotic or embolic events such as a stroke and transient ischemic attack within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ NCI CTCAE v3.0 Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ NCI CTCAE v3.0 Grade 3 within 4 weeks of first dose of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Methodist Cancer Center, Omaha, Nebraska
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Background] Spigel DR, Hainsworth JD, Burris HA 3rd, Molthrop DC, Peacock N, Kommor M, Vazquez ER, Greco FA, Yardley DA. A pilot study of adjuvant doxorubicin and cyclophosphamide followed by paclitaxel and sorafenib in women with node-positive or high-risk early-stage breast cancer. Clin Adv Hematol Oncol. 2011 Apr;9(4):280-6. PMID 21558987
- See also: Related Info — http://www.clinicaladvances.com/index.php/our_publications/hem_onc-article/1980/

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib: All patients received doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2 (AC) both administered intravenously day 1 every 3 weeks for four cycles, followed by paclitaxel 175 mg/m2 intravenously day 1 every 3 weeks for four cycles or 80 mg/m2 for twelve weeks (physician discretion), combined with sorafenib 400 mg orally twice daily. Sorafenib was held during radiation therapy where indicated and resumed once completed. Sorafenib was continued for a total of 12 months and in combination with adjuvant hormonal therapy where indicated.
Period: Overall Study
Arm/Group | Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib
Started | 45
Completed | 16
Not Completed | 29
Not completed — Adverse Event | 21
Not completed — Physician Decision | 8

BASELINE CHARACTERISTICS:
Groups:
- Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib: Doxorubicin 60mg/m2 IV, Cyclophosphamide 600mg/m2 IV every 3 weeks for a total of 12 weeks followed by 12 weeks of paclitaxel (either 175mg/m2 IV every three weeks or 80mg/m2 IV weekly) and sorafenib 400mg twice daily by mouth (up to a maximum of 1 year).
Arm/Group | Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib
Number analyzed (Participants) | 45
Age Continuous [Median (Full Range); unit: years] | 54 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability of Protocol Treatment, Defined as the Percentage of Patients Experiencing Severe or Life-threatening Side Effects Per CTCAE Version 3.0.
Time Frame: 18 Months
Measure: Number; unit: percentage of patients
Arm/Group | Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib
Number analyzed (Participants) | 45
percentage of patients | 40

ADVERSE EVENTS:
Arm/Group | Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib
Serious Adverse Events (participants affected / at risk) | 7/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib (N=45)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Infection - pneumonia (Infections and infestations) | 1 (1)
Abcess of Bartholin's cyst (Reproductive system and breast disorders) | 1 (1)
Hemmorhage - GI (Gastrointestinal disorders) | 1 (1)
Infection - Streptococcus (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ventricular arrhythmia - left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin/Cyclophosphamide Then Paclitaxel/Sorafenib (N=45)
Pain - Abdomen (Gastrointestinal disorders) | 10 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 31 (158)
Anorexia (Gastrointestinal disorders) | 11 (39)
Mood Alteration - Anxiety (Psychiatric disorders) | 8 (26)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 19 (47)
Superventricular arrhythmia - Atrial Fibrillation (Cardiac disorders) | 7 (12)
Blurred Vision (Eye disorders) | 5 (14)
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 14 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (19)
Mood Alteration - Depression (Psychiatric disorders) | 5 (18)
Diarrhea (Gastrointestinal disorders) | 17 (55)
Dizziness (Nervous system disorders) | 6 (6)
Dry Mouth (Gastrointestinal disorders) | 3 (8)
Taste Alteration (Gastrointestinal disorders) | 3 (4)
Heartburn (Gastrointestinal disorders) | 4 (10)
Dysphagia (Gastrointestinal disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (23)
Edema (Blood and lymphatic system disorders) | 4 (13)
Hemorrhage Pulmonary - Nose (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Esophagitis (Gastrointestinal disorders) | 3 (11)
Fatigue (General disorders) | 40 (228)
Fever (General disorders) | 11 (15)
Hand-Foot (Skin and subcutaneous tissue disorders) | 13 (54)
Hemoglobin (Blood and lymphatic system disorders) | 42 (169)
Hot Flashes (Endocrine disorders) | 8 (13)
Hyperglycemia (Endocrine disorders) | 5 (27)
Hypertension (Cardiac disorders) | 9 (22)
Hypokalemia (Endocrine disorders) | 4 (5)
Infection - URI (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Infection (Infections and infestations) | 7 (10) — Without Grade 3/4 ANC
Insomnia (General disorders) | 7 (10)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 4 (5)
Watery Eye (Eye disorders) | 4 (28)
Leukocytes (Blood and lymphatic system disorders) | 37 (161)
Mouth Sore (Gastrointestinal disorders) | 4 (9)
Muscositis - Oral Cavity (Gastrointestinal disorders) | 20 (55)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 22 (47)
Nail Changes (Skin and subcutaneous tissue disorders) | 4 (15)
Nausea (Gastrointestinal disorders) | 40 (125)
Neuropathy - Peripheral (Nervous system disorders) | 4 (23)
Neuropathy - Sensory (Nervous system disorders) | 28 (89)
Neutrophils (Blood and lymphatic system disorders) | 34 (111)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 10 (16)
Pain - Ear (Ear and labyrinth disorders) | 3 (3)
Pain - Headache (General disorders) | 9 (12)
Infection - Pharynx (Infections and infestations) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 17 (37)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (17)
Pruritis (Skin and subcutaneous tissue disorders) | 9 (16)
Rash (Skin and subcutaneous tissue disorders) | 26 (88)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 (14)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (6)
Pain - Throat (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Tachycardia (Cardiac disorders) | 8 (16)
Taste Alteration (Gastrointestinal disorders) | 11 (58)
Vomiting (Gastrointestinal disorders) | 21 (53)
Weakness (General disorders) | 3 (12)
Weight Loss (General disorders) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.